CLINICAL TRIAL: NCT01050062
Title: Post Marketing Surveillance on Long Drug Use of Micombi Combination Tablets in Patients With Hypertension
Brief Title: Post-Marketing Surveillance of Micombi Tablets Survey on the Long-term Use
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: 502.542
Record Dates: First submitted 2009-12-24; First posted 2010-01-15 (Estimated); Results first posted 2013-01-30 (Estimated); Last update posted 2014-05-01 (Estimated); Status verified 2014-04

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Telmisartan; Hydrochlorothiazide

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Micombi® Combination Tablet AP
  Interventions: Drug: Telmisartan 40mg; Drug: Hydrochlorothiazide 12.5mg
- Micombi® Combination Tablet BP
  Interventions: Drug: Telmisartan 80mg; Drug: Hydrochlorothiazide 12.5mg

INTERVENTIONS:
Drug: Telmisartan 80mg — Combination tablet
  Groups: Micombi® Combination Tablet BP
Drug: Telmisartan 40mg — Combination tablet
  Groups: Micombi® Combination Tablet AP
Drug: Hydrochlorothiazide 12.5mg — Combination tablet

SUMMARY:
The survey is conducted to collect safety and effectiveness information in Hypertensive patients treated with Micombi Tablets on the long term use in daily clinical settings in Japan.

ELIGIBILITY:
Inclusion criteria:

Hypertensive patients who have never taken Micombi Tablets.

Exclusion criteria:

None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 1000
Sampling Method: Non-Probability Sample
Enrollment: 1452 (Actual)
Dates: Start 2010-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (314):
- Japan (314):
  - Boehringer Ingelheim Investigational Site 111, Ageo
  - Boehringer Ingelheim Investigational Site 209, Aisho-cho
  - Boehringer Ingelheim Investigational Site 22, Aizubange-machi
  - Boehringer Ingelheim Investigational Site 234, Akashi
  - Boehringer Ingelheim Investigational Site 78, Akiruno
  - Boehringer Ingelheim Investigational Site 79, Akishima
  - Boehringer Ingelheim Investigational Site 235, Akō
  - Boehringer Ingelheim Investigational Site 288, Akune
  - Boehringer Ingelheim Investigational Site 236, Amagasaki
  - Boehringer Ingelheim Investigational Site 237, Amagasaki
  - Boehringer Ingelheim Investigational Site 280, Anan
  - Boehringer Ingelheim Investigational Site 160, Anjo
  - Boehringer Ingelheim Investigational Site 1, Asahikawa
  - Boehringer Ingelheim Investigational Site 51, Ashikaga
  - Boehringer Ingelheim Investigational Site 140, Atsugi
  - Boehringer Ingelheim Investigational Site 58, Azumino
  - Boehringer Ingelheim Investigational Site 128, Chiba
  - Boehringer Ingelheim Investigational Site 138, Chiba
  - Boehringer Ingelheim Investigational Site 141, Chigasaki
  - Boehringer Ingelheim Investigational Site 299, Chikujo-machi
  - Boehringer Ingelheim Investigational Site 44, Chikusei
  - Boehringer Ingelheim Investigational Site 80, Chōfu
  - Boehringer Ingelheim Investigational Site 311, Ebino
  - Boehringer Ingelheim Investigational Site 257, Fuchū
  - Boehringer Ingelheim Investigational Site 71, Fuefuki
  - Boehringer Ingelheim Investigational Site 179, Fujieda
  - Boehringer Ingelheim Investigational Site 211, Fujiidera
  - Boehringer Ingelheim Investigational Site 112, Fukaya
  - Boehringer Ingelheim Investigational Site 206, Fukui
  - Boehringer Ingelheim Investigational Site 300, Fukuoka
  - Boehringer Ingelheim Investigational Site 301, Fukuoka
  - Boehringer Ingelheim Investigational Site 302, Fukuoka
  - Boehringer Ingelheim Investigational Site 303, Fukuoka
  - Boehringer Ingelheim Investigational Site 180, Fukuroi
  - Boehringer Ingelheim Investigational Site 23, Fukushima
  - Boehringer Ingelheim Investigational Site 258, Fukuyama
  - Boehringer Ingelheim Investigational Site 129, Funabashi
  - Boehringer Ingelheim Investigational Site 47, Funaishikawa
  - Boehringer Ingelheim Investigational Site 174, Gifu
  - Boehringer Ingelheim Investigational Site 175, Gifu
  - Boehringer Ingelheim Investigational Site 42, Gonohe-machi
  - Boehringer Ingelheim Investigational Site 113, Gyōda
  - Boehringer Ingelheim Investigational Site 212, Habikino
  - Boehringer Ingelheim Investigational Site 81, Hachiōji
  - Boehringer Ingelheim Investigational Site 82, Hachiōji
  - Boehringer Ingelheim Investigational Site 193, Hakusan
  - Boehringer Ingelheim Investigational Site 181, Hamamatsu
  - Boehringer Ingelheim Investigational Site 247, Hashimoto
  - Boehringer Ingelheim Investigational Site 142, Hatano
  - Boehringer Ingelheim Investigational Site 259, Hatsukaichi
  - Boehringer Ingelheim Investigational Site 114, Higashi-Matsuyama
  - Boehringer Ingelheim Investigational Site 276, Higashikagawa
  - Boehringer Ingelheim Investigational Site 83, Higashikurume
  - Boehringer Ingelheim Investigational Site 213, Higashiosaka
  - Boehringer Ingelheim Investigational Site 84, Hino
  - Boehringer Ingelheim Investigational Site 43, Hirosaki
  - Boehringer Ingelheim Investigational Site 260, Hiroshima
  - Boehringer Ingelheim Investigational Site 261, Hiroshima
  - Boehringer Ingelheim Investigational Site 262, Hiroshima
  - Boehringer Ingelheim Investigational Site 263, Hiroshima
  - Boehringer Ingelheim Investigational Site 45, Hitachi-Naka
  - Boehringer Ingelheim Investigational Site 72, Hokuto
  - Boehringer Ingelheim Investigational Site 266, Hōfu
  - Boehringer Ingelheim Investigational Site 249, Ibara
  - Boehringer Ingelheim Investigational Site 214, Ibaraki
  - Boehringer Ingelheim Investigational Site 215, Ibaraki
  - Boehringer Ingelheim Investigational Site 130, Ichikawa
  - Boehringer Ingelheim Investigational Site 161, Ichinomiya
  - Boehringer Ingelheim Investigational Site 18, Ichinoseki
  - Boehringer Ingelheim Investigational Site 19, Ichinoseki
  - Boehringer Ingelheim Investigational Site 59, Ina
  - Boehringer Ingelheim Investigational Site 289, Isa
  - Boehringer Ingelheim Investigational Site 187, Ise
  - Boehringer Ingelheim Investigational Site 74, Isesaki
  - Boehringer Ingelheim Investigational Site 182, Itō
  - Boehringer Ingelheim Investigational Site 52, Iwafune-machi
  - Boehringer Ingelheim Investigational Site 24, Iwaki
  - Boehringer Ingelheim Investigational Site 162, Iwakura
  - Boehringer Ingelheim Investigational Site 216, Izumisano
  - Boehringer Ingelheim Investigational Site 194, Kaga
  - Boehringer Ingelheim Investigational Site 290, Kagoshima
  - Boehringer Ingelheim Investigational Site 73, Kai
  - Boehringer Ingelheim Investigational Site 195, Kanazawa
  - Boehringer Ingelheim Investigational Site 53, Kanuma
  - Boehringer Ingelheim Investigational Site 163, Kariya
  - Boehringer Ingelheim Investigational Site 238, Kasai
  - Boehringer Ingelheim Investigational Site 164, Kasugai
  - Boehringer Ingelheim Investigational Site 115, Kasukabe
  - Boehringer Ingelheim Investigational Site 217, Kawachi-Nagano
  - Boehringer Ingelheim Investigational Site 116, Kawaguchi
  - Boehringer Ingelheim Investigational Site 117, Kawaguchi
  - Boehringer Ingelheim Investigational Site 231, Kawaichō
  - Boehringer Ingelheim Investigational Site 143, Kawasaki
  - Boehringer Ingelheim Investigational Site 144, Kawasaki
  - Boehringer Ingelheim Investigational Site 145, Kawasaki
  - Boehringer Ingelheim Investigational Site 296, Kawatana-cho
  - Boehringer Ingelheim Investigational Site 40, Kazuno
  - Boehringer Ingelheim Investigational Site 29, Kesennuma
  - Boehringer Ingelheim Investigational Site 131, Kisarazu
  - Boehringer Ingelheim Investigational Site 2, Kitahiroshima
  - Boehringer Ingelheim Investigational Site 304, Kitakyushu
  - Boehringer Ingelheim Investigational Site 305, Kitakyushu
  - Boehringer Ingelheim Investigational Site 306, Kitakyushu
  - Boehringer Ingelheim Investigational Site 239, Kobe
  - Boehringer Ingelheim Investigational Site 240, Kobe
  - Boehringer Ingelheim Investigational Site 241, Kobe
  - Boehringer Ingelheim Investigational Site 242, Kobe
  - Boehringer Ingelheim Investigational Site 118, Koshigaya
  - Boehringer Ingelheim Investigational Site 277, Kotohira
  - Boehringer Ingelheim Investigational Site 25, Kōriyama
  - Boehringer Ingelheim Investigational Site 119, Kumagaya
  - Boehringer Ingelheim Investigational Site 291, Kumamoto
  - Boehringer Ingelheim Investigational Site 292, Kumamoto
  - Boehringer Ingelheim Investigational Site 284, Kunisaki
  - Boehringer Ingelheim Investigational Site 250, Kurashiki
  - Boehringer Ingelheim Investigational Site 264, Kure
  - Boehringer Ingelheim Investigational Site 265, Kure
  - Boehringer Ingelheim Investigational Site 285, Kusu-machi
  - Boehringer Ingelheim Investigational Site 197, Kyoto
  - Boehringer Ingelheim Investigational Site 198, Kyoto
  - Boehringer Ingelheim Investigational Site 199, Kyoto
  - Boehringer Ingelheim Investigational Site 200, Kyoto
  - Boehringer Ingelheim Investigational Site 85, Machida
  - Boehringer Ingelheim Investigational Site 307, Maebaru
  - Boehringer Ingelheim Investigational Site 146, Matsuda-machi
  - Boehringer Ingelheim Investigational Site 132, Matsudo
  - Boehringer Ingelheim Investigational Site 60, Matsumoto
  - Boehringer Ingelheim Investigational Site 61, Matsumoto
  - Boehringer Ingelheim Investigational Site 272, Matsuyama
  - Boehringer Ingelheim Investigational Site 273, Matsuyama
  - Boehringer Ingelheim Investigational Site 188, Matsuzaka
  - Boehringer Ingelheim Investigational Site 293, Minamata
  - Boehringer Ingelheim Investigational Site 30, Minamisanriku
  - Boehringer Ingelheim Investigational Site 218, Minoo
  - Boehringer Ingelheim Investigational Site 46, Mito
  - Boehringer Ingelheim Investigational Site 312, Miyazaki
  - Boehringer Ingelheim Investigational Site 133, Mobara
  - Boehringer Ingelheim Investigational Site 20, Morioka
  - Boehringer Ingelheim Investigational Site 26, Motomiya
  - Boehringer Ingelheim Investigational Site 3, Mukawa-cho
  - Boehringer Ingelheim Investigational Site 86, Musashino
  - Boehringer Ingelheim Investigational Site 62, Nagano
  - Boehringer Ingelheim Investigational Site 63, Nagano
  - Boehringer Ingelheim Investigational Site 297, Nagasaki
  - Boehringer Ingelheim Investigational Site 165, Nagoya
  - Boehringer Ingelheim Investigational Site 166, Nagoya
  - Boehringer Ingelheim Investigational Site 167, Nagoya
  - Boehringer Ingelheim Investigational Site 168, Nagoya
  - Boehringer Ingelheim Investigational Site 192, Nagoya
  - Boehringer Ingelheim Investigational Site 314, Naha
  - Boehringer Ingelheim Investigational Site 41, Nakadōri
  - Boehringer Ingelheim Investigational Site 54, Nakagawamachi
  - Boehringer Ingelheim Investigational Site 176, Nakatsugawa
  - Boehringer Ingelheim Investigational Site 196, Nanao
  - Boehringer Ingelheim Investigational Site 278, Nankoku
  - Boehringer Ingelheim Investigational Site 232, Nara
  - Boehringer Ingelheim Investigational Site 31, Natori
  - Boehringer Ingelheim Investigational Site 4, Nayoro
  - Boehringer Ingelheim Investigational Site 313, Nichinan
  - Boehringer Ingelheim Investigational Site 65, Niigata
  - Boehringer Ingelheim Investigational Site 66, Niigata
  - Boehringer Ingelheim Investigational Site 147, Ninomiya-machi
  - Boehringer Ingelheim Investigational Site 243, Nishinomiya
  - Boehringer Ingelheim Investigational Site 244, Nishinomiya
  - Boehringer Ingelheim Investigational Site 169, Nishio
  - Boehringer Ingelheim Investigational Site 87, Nishitōkyō
  - Boehringer Ingelheim Investigational Site 5, Obihiro
  - Boehringer Ingelheim Investigational Site 255, Oda
  - Boehringer Ingelheim Investigational Site 189, Odai-cho
  - Boehringer Ingelheim Investigational Site 148, Odawara
  - Boehringer Ingelheim Investigational Site 294, Ogi
  - Boehringer Ingelheim Investigational Site 251, Okayama
  - Boehringer Ingelheim Investigational Site 252, Okayama
  - Boehringer Ingelheim Investigational Site 253, Okayama
  - Boehringer Ingelheim Investigational Site 308, Omuta
  - Boehringer Ingelheim Investigational Site 309, Omuta
  - Boehringer Ingelheim Investigational Site 219, Osaka
  - Boehringer Ingelheim Investigational Site 220, Osaka
  - Boehringer Ingelheim Investigational Site 221, Osaka
  - Boehringer Ingelheim Investigational Site 222, Osaka
  - Boehringer Ingelheim Investigational Site 223, Osaka
  - Boehringer Ingelheim Investigational Site 224, Osaka
  - Boehringer Ingelheim Investigational Site 225, Osaka
  - Boehringer Ingelheim Investigational Site 226, Osaka
  - Boehringer Ingelheim Investigational Site 6, Otaru
  - Boehringer Ingelheim Investigational Site 55, Oyama
  - Boehringer Ingelheim Investigational Site 16, Ōdate
  - Boehringer Ingelheim Investigational Site 286, Ōita
  - Boehringer Ingelheim Investigational Site 287, Ōita
  - Boehringer Ingelheim Investigational Site 21, Ōshū
  - Boehringer Ingelheim Investigational Site 210, Ōtsu
  - Boehringer Ingelheim Investigational Site 75, Ōuramachi
  - Boehringer Ingelheim Investigational Site 67, Sado
  - Boehringer Ingelheim Investigational Site 149, Sagamihara
  - Boehringer Ingelheim Investigational Site 150, Sagamihara
  - Boehringer Ingelheim Investigational Site 274, Saijō
  - Boehringer Ingelheim Investigational Site 120, Saitama
  - Boehringer Ingelheim Investigational Site 121, Saitama
  - Boehringer Ingelheim Investigational Site 122, Saitama
  - Boehringer Ingelheim Investigational Site 227, Sakai
  - Boehringer Ingelheim Investigational Site 228, Sakai
  - Boehringer Ingelheim Investigational Site 229, Sakai
  - Boehringer Ingelheim Investigational Site 39, Sakata
  - Boehringer Ingelheim Investigational Site 134, Sakura
  - Boehringer Ingelheim Investigational Site 68, Sanjō
  - Boehringer Ingelheim Investigational Site 135, Sanmu
  - Boehringer Ingelheim Investigational Site 267, Sanyōonoda
  - Boehringer Ingelheim Investigational Site 268, Sanyōonoda
  - Boehringer Ingelheim Investigational Site 10, Sapporo
  - Boehringer Ingelheim Investigational Site 11, Sapporo
  - Boehringer Ingelheim Investigational Site 12, Sapporo
  - Boehringer Ingelheim Investigational Site 7, Sapporo
  - Boehringer Ingelheim Investigational Site 8, Sapporo
  - Boehringer Ingelheim Investigational Site 9, Sapporo
  - Boehringer Ingelheim Investigational Site 298, Sasebo
  - Boehringer Ingelheim Investigational Site 123, Satte
  - Boehringer Ingelheim Investigational Site 124, Sayama
  - Boehringer Ingelheim Investigational Site 32, Sendai
  - Boehringer Ingelheim Investigational Site 33, Sendai
  - Boehringer Ingelheim Investigational Site 34, Sendai
  - Boehringer Ingelheim Investigational Site 35, Sendai
  - Boehringer Ingelheim Investigational Site 36, Sendai
  - Boehringer Ingelheim Investigational Site 37, Sendai
  - Boehringer Ingelheim Investigational Site 69, Shibata
  - Boehringer Ingelheim Investigational Site 13, Shibetsu
  - Boehringer Ingelheim Investigational Site 125, Shiki
  - Boehringer Ingelheim Investigational Site 279, Shimanto
  - Boehringer Ingelheim Investigational Site 310, Shime-machi
  - Boehringer Ingelheim Investigational Site 183, Shimoda
  - Boehringer Ingelheim Investigational Site 248, Shingū
  - Boehringer Ingelheim Investigational Site 38, Shiraishi
  - Boehringer Ingelheim Investigational Site 136, Shiroi
  - Boehringer Ingelheim Investigational Site 184, Shizuoka
  - Boehringer Ingelheim Investigational Site 185, Shizuoka
  - Boehringer Ingelheim Investigational Site 269, Shūnan
  - Boehringer Ingelheim Investigational Site 126, Sōka
  - Boehringer Ingelheim Investigational Site 27, Sukagawa
  - Boehringer Ingelheim Investigational Site 190, Suzuka
  - Boehringer Ingelheim Investigational Site 88, Tachikawa
  - Boehringer Ingelheim Investigational Site 203, Takaoka
  - Boehringer Ingelheim Investigational Site 204, Takaoka
  - Boehringer Ingelheim Investigational Site 245, Takarazuka
  - Boehringer Ingelheim Investigational Site 76, Takasaki
  - Boehringer Ingelheim Investigational Site 77, Takasaki
  - Boehringer Ingelheim Investigational Site 177, Takayama
  - Boehringer Ingelheim Investigational Site 246, Tatsuno
  - Boehringer Ingelheim Investigational Site 170, Tokoname
  - Boehringer Ingelheim Investigational Site 127, Tokorozawa
  - Boehringer Ingelheim Investigational Site 281, Tokushima
  - Boehringer Ingelheim Investigational Site 282, Tokushima
  - Boehringer Ingelheim Investigational Site 89, Tokyo Adachi-ku
  - Boehringer Ingelheim Investigational Site 90, Tokyo Adachi-ku
  - Boehringer Ingelheim Investigational Site 102, Tokyo Bunkyo-ku
  - Boehringer Ingelheim Investigational Site 91, Tokyo Chiyoda-ku
  - Boehringer Ingelheim Investigational Site 92, Tokyo Chiyoda-ku
  - Boehringer Ingelheim Investigational Site 93, Tokyo Kita-ku
  - Boehringer Ingelheim Investigational Site 94, Tokyo Koto-ku
  - Boehringer Ingelheim Investigational Site 95, Tokyo Meguro-ku
  - Boehringer Ingelheim Investigational Site 96, Tokyo Meguro-ku
  - Boehringer Ingelheim Investigational Site 97, Tokyo Nerima-ku
  - Boehringer Ingelheim Investigational Site 98, Tokyo Ota-ku
  - Boehringer Ingelheim Investigational Site 99, Tokyo Ota-ku
  - Boehringer Ingelheim Investigational Site 100, Tokyo Setagaya-ku
  - Boehringer Ingelheim Investigational Site 101, Tokyo Setagaya-ku
  - Boehringer Ingelheim Investigational Site 103, Tokyo Shibuya-ku
  - Boehringer Ingelheim Investigational Site 104, Tokyo Shinagawa-ku
  - Boehringer Ingelheim Investigational Site 105, Tokyo Shinagawa-ku
  - Boehringer Ingelheim Investigational Site 106, Tokyo Shinagawa-ku
  - Boehringer Ingelheim Investigational Site 107, Tokyo Shinjuku-ku
  - Boehringer Ingelheim Investigational Site 108, Tokyo Suginami-ku
  - Boehringer Ingelheim Investigational Site 109, Tokyo Sumida-ku
  - Boehringer Ingelheim Investigational Site 110, Tokyo Toshima-ku
  - Boehringer Ingelheim Investigational Site 14, Tomakomai
  - Boehringer Ingelheim Investigational Site 28, Tomioka
  - Boehringer Ingelheim Investigational Site 295, Tosu
  - Boehringer Ingelheim Investigational Site 270, Tottori
  - Boehringer Ingelheim Investigational Site 15, Toyako-machi
  - Boehringer Ingelheim Investigational Site 205, Toyama
  - Boehringer Ingelheim Investigational Site 171, Toyohashi
  - Boehringer Ingelheim Investigational Site 172, Toyokawa
  - Boehringer Ingelheim Investigational Site 230, Toyonaka
  - Boehringer Ingelheim Investigational Site 173, Toyota
  - Boehringer Ingelheim Investigational Site 70, Tōkamachi
  - Boehringer Ingelheim Investigational Site 49, Tsuchiura
  - Boehringer Ingelheim Investigational Site 207, Tsuruga
  - Boehringer Ingelheim Investigational Site 208, Tsuruga
  - Boehringer Ingelheim Investigational Site 283, Tsurugi-cho
  - Boehringer Ingelheim Investigational Site 254, Tsuyama
  - Boehringer Ingelheim Investigational Site 64, Ueda
  - Boehringer Ingelheim Investigational Site 201, Uji
  - Boehringer Ingelheim Investigational Site 48, Ushiku
  - Boehringer Ingelheim Investigational Site 56, Utsunomiya
  - Boehringer Ingelheim Investigational Site 57, Utsunomiya
  - Boehringer Ingelheim Investigational Site 275, Uwajima
  - Boehringer Ingelheim Investigational Site 137, Yachimata
  - Boehringer Ingelheim Investigational Site 186, Yaizu
  - Boehringer Ingelheim Investigational Site 178, Yamagata
  - Boehringer Ingelheim Investigational Site 151, Yamato
  - Boehringer Ingelheim Investigational Site 233, Yamatokooriyama
  - Boehringer Ingelheim Investigational Site 191, Yokkaichi
  - Boehringer Ingelheim Investigational Site 152, Yokohama
  - Boehringer Ingelheim Investigational Site 153, Yokohama
  - Boehringer Ingelheim Investigational Site 154, Yokohama
  - Boehringer Ingelheim Investigational Site 155, Yokohama
  - Boehringer Ingelheim Investigational Site 156, Yokohama
  - Boehringer Ingelheim Investigational Site 157, Yokohama
  - Boehringer Ingelheim Investigational Site 158, Yokohama
  - Boehringer Ingelheim Investigational Site 159, Yokosuka
  - Boehringer Ingelheim Investigational Site 271, Yonago
  - Boehringer Ingelheim Investigational Site 202, Yosano-cho
  - Boehringer Ingelheim Investigational Site 256, Yoshika-cho
  - Boehringer Ingelheim Investigational Site 139, Yotsukaidō
  - Boehringer Ingelheim Investigational Site 17, Yurihonjō
  - Boehringer Ingelheim Investigational Site 50, Yūki

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 1452 patients were enrolled. Of these patients, the CRFs of 9 patients were uncollected by reason of institution, and the 18 patients which were no information including safety due to no visit after enrolled. Then, total 1425 patients were observed in the survey.
Groups:
- Combination Tablet AP: Fix dose combination tablets of telmisartan 40mg and hydrochlorothiazide 12.5mg
- Combination Tablet BP: Fix dose combination tablets of telmisartan 80mg and hydrochlorothiazide 12.5mg
Period: Overall Study
Arm/Group | Combination Tablet AP | Combination Tablet BP
Started | 1070 | 355
Completed | 799 | 243
Not Completed | 271 | 112
Not completed — Adverse Event | 75 | 22
Not completed — Lost to Follow-up | 83 | 35
Not completed — Lack of Efficacy | 22 | 35
Not completed — Physician Decision | 74 | 9
Not completed — Others | 17 | 11

BASELINE CHARACTERISTICS:
Population: The 18 patients which had no information including safety due to no visit after enrolled, were excluded from the safety analysis, 1,425 patients were included in the safety set.
Groups:
- Total: Total of all reporting groups
Arm/Group | Combination Tablet AP | Combination Tablet BP | Total
Number analyzed (Participants) | 1070 | 355 | 1425
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.6 (12.0) | 69.8 (12.5) | 68.9 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 570 | 186 | 756
  Male | 500 | 169 | 669

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Adverse Events (AEs)
Description: The number of patient with any AEs, patients with drug-related AEs
Time Frame: Week 52
Population: The all treated patients, 18 patients which were no information including safety due to no visit after enrolled. Then, total 1425 patients were observed in the survey
Measure: Number; unit: Patients
Groups:
- Total: Fix dose combination tablets of telmisartan 40/80mg and hydrochlorothiazide 12.5mg
Arm/Group | Combination Tablet AP | Combination Tablet BP | Total
Number analyzed (Participants) | 1070 | 355 | 1425
Patients
  patient with any AEs | 221 | 72 | 293
  patients with drug-related AEs | 154 | 46 | 200

2. Secondary Outcome: Systolic Blood Pressure (SBP)
Description: SBP is observed at Week 0 and Week 52. The change of SBP from Week 0 to Week 52 is calculated.
Time Frame: Week 0 and Week 52
Population: The 13 patients which no efficacy information, were excluding from safety set, 1412 patients were included in efficacy set.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Combination Tablet AP | Combination Tablet BP | Total
Number analyzed (Participants) | 1060 | 352 | 1412
mmHg
  Week 0 | 152.9 (18.3) | 155.4 (18.7) | 153.5 (18.4)
  Week 52 | 132.2 (15.1) | 134.7 (15.5) | 132.8 (15.2)
  Change from Week 0 to Week 52 | -20.7 (18.8) | -20.7 (21.5) | -20.7 (19.5)

3. Secondary Outcome: Diastolic Blood Pressure (DBP)
Description: DBP is observed at Week 0 and Week 52. The change of DBP from Week 0 to Week 52 is calculated.
Time Frame: Week 0 and Week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Combination Tablet AP | Combination Tablet BP | Total
Number analyzed (Participants) | 1060 | 352 | 1412
mmHg
  Week 0 | 84.7 (13.0) | 84.6 (12.8) | 84.7 (13.0)
  Week 52 | 75.2 (10.9) | 75.5 (11.2) | 75.3 (11.0)
  Change from Week 0 to Week 52 | -9.5 (11.6) | -9.1 (13.9) | -9.4 (12.2)

4. Secondary Outcome: Target Blood Pressure Achievement Rate
Description: The proportion of the patients with target blood pressure in 52 weeks administrative period. Target blood pressure is defined as 'Guidelines for the management of hypertension (JSH2009)': less than 140/90 (SBP/DBP) mmHg for >= 65 years old or cerebrovascular disorder patient; less than 130/80 in diabetes, chronic kidney disease or myocardial infarction patient; less than 130/85 mmHg for others patient.
Time Frame: Week 52
Population: as for outcome 2
Measure: Number; unit: Percentage of patients
Arm/Group | Combination Tablet AP | Combination Tablet BP | Total
Number analyzed (Participants) | 1060 | 352 | 1412
Percentage of patients | 52.9 | 43.2 | 50.5

5. Secondary Outcome: Blood Pressure Normalised Rate
Description: The proportion of the patients with normalized blood pressure in 52 weeks on administrative period. Normalized blood pressure is defined less than 140/90 (SBP/DBP) mmHg according to JSH2009
Time Frame: Week 52
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Combination Tablet AP | Combination Tablet BP | Total
Number analyzed (Participants) | 1060 | 352 | 1412
percentage of participants | 70.7 | 61.1 | 68.3

ADVERSE EVENTS:
Time Frame: 52 weeks
Arm/Group | Combination Tablet Ap | Combination Tablet BP | Total
Serious Adverse Events (participants affected / at risk) | 25/1070 | 12/355 | 37/1425
Other Adverse Events (participants affected / at risk) | 0/1070 | 0/355 | 0/1425
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Combination Tablet Ap (N=1070) | Combination Tablet BP (N=355) | Total (N=1425)
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 1
Angina pectoris (Cardiac disorders) | 1 | 0 | 1
Angina unstable (Cardiac disorders) | 0 | 1 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 1
Sick sinus syndrome (Cardiac disorders) | 1 | 0 | 1
Autoimmune pancreatitis (Gastrointestinal disorders) | 1 | 0 | 1
Death (General disorders) | 0 | 1 | 1
Cholangitis acute (Hepatobiliary disorders) | 1 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 2 | 0 | 2
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 1 | 1
Gastroenteritis (Infections and infestations) | 1 | 0 | 1
Arthritis bacterial (Infections and infestations) | 0 | 1 | 1
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 1
Pneumocystis jiroveci pneumonia (Infections and infestations) | 1 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 1 | 3
Hypophagia (Metabolism and nutrition disorders) | 1 | 0 | 1
Mixed connective tissue disease (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Cerebral infarction (Nervous system disorders) | 3 | 1 | 4
Cerebrovascular disorder (Nervous system disorders) | 0 | 1 | 1
Loss of consciousness (Nervous system disorders) | 1 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 1
Completed suicide (Psychiatric disorders) | 1 | 0 | 1
Calculus urinary (Renal and urinary disorders) | 0 | 1 | 1
Renal failure chronic (Renal and urinary disorders) | 1 | 1 | 2
Renal impairment (Renal and urinary disorders) | 1 | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes